CLINICAL TRIAL: NCT07144605
Title: Comparison of the Long-Term Success of Different CAD-CAM Blocks Used as Indirect Restorations in Molar Incisor Hypomineralized Teeth: A Split Mouth Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Halenur Altan, Professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NecmettinEU05
Record Dates: First submitted 2025-07-15; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Molar Hypomineralization, Incisor
Keywords: CAD-CAM, Indirect restorations; Molar Incisor Hypomineralization; MIH
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Intervention Model Description: In our study, treatment was planned for moderately affected teeth according to the MIH Severity Index. The study was designed as a prospective, randomized, split-mouth trial. Group randomization was performed using the sealed envelope technique. In the same patient, VOCO GrandioBloc (VOCO GmbH, Cuxhaven, Germany) was applied to one tooth, while a GC Initial lithium disilicate block was applied to the symmetrical contralateral tooth.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Voco Grandio blocs(Grandio Blocs (R) VOCO) (Experimental): Nanohybrid ceramic blocks, indirect restorative materials
  Interventions: Other: CAD-CAM, indirect restorations
- GC INITIAL LiSi Blocs (GC AMERICA INC. USA) (Experimental): Glass ceramic blocks, indirect restorative materials
  Interventions: Other: CAD-CAM, indirect restorations

INTERVENTIONS:
Other: CAD-CAM, indirect restorations — Indirect restorations that we think will last longer than traditional filling materials in teeth with molar hypomineralization.

SUMMARY:
This study is about the long-term survival success of different, externally prepared fillings (Indirect restoration, CAD-CAM blocks) used in teeth with reduced mineral structure, namely Molar Incisor Hypomineralization (MIH), which is called chalk teeth in children.

DETAILED DESCRIPTION:
The aim of this study was to comparatively evaluate the long-term survival times and clinical success of nano-ceramic hybrid CAD-CAM blocks, Grandio Blocs (R) (VOCO), and glass-ceramic blocks, GC INITIAL LiSi (GC AMERICA INC. USA), according to USPHS criteria, after pulpal treatment in mandibular teeth with bilateral moderate molar incisor hypomineralization.

ELIGIBILITY:
Inclusion Criteria:8-15 years old

* Systemically healthy
* Cooperative (Frankl 3-4)
* Diagnosed with MIH for at least one permanent tooth
* Symmetrical mandibular molars that fit the middle MIH classification (teeth with a tooth score of 7-9 in MIHSI)
* Teeth without indication for root canal treatment
* Teeth without percussion, abscess and fistula formation
* Without periapical lesions
* With post-eruption enamel fractures in the relevant teeth
* Without mobility and pathological gingival pockets
* Patients who agreed to participate in the study.

Exclusion Criteria:Teeth that are suitable for mild and severe classification

* Non-cooperative (Frankl 1 and Frankl 2)
* Teeth with extraction indication
* Teeth that require root canal treatment
* Teeth with periapical lesions, abscesses and fistula formation
* Patients with mobility and pathological gingival pockets

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
the clinical status of the restorations | up to 6 months after intervention
  The restorations were clinically evaluated in the oral cavity using the USPHS index.
the status of the periapical tissues | Up to the 6th months
  The periapical tissue status was assessed according to the Periapical Index (PAI).

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The participants don't want to share the individual information about study.

REFERENCES:
- See also: https://link.springer.com/article/10.1007/s10266-023-00841-w — https://link.springer.com/article/10.1007/s10266-023-00841-w